CLINICAL TRIAL: NCT02953665
Title: A Phase II, Randomized, Double-blinded, Placebo-controlled Trial of Liraglutide in Parkinson's Disease
Brief Title: Safety and Efficacy of Liraglutide in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Cure Parkinson's (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Michele Tagliati, MD, Director, Movement Disorders, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1173-0106
Record Dates: First submitted 2016-10-21; First posted 2016-11-03 (Estimated); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease, Liraglutide; Antidiabetic agents; GLP-1 agonists; Insulin resistance
MeSH Terms: conditions — Parkinson Disease; Insulin Resistance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Active Comparator): Liraglutide 6 mg/ml (Novo Nordisk A/S) will be self-administered subcutaneously once daily at a maximum dose of 1.8 mg after a 2 week titration schedule.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo will be self-administered subcutaneously once daily according to the same schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide 6 mg/ml once daily at a maximum dose of 1.8 mg
  Other Names: Victoza; Saxenda
  Arms: Liraglutide
Drug: Placebo — Placebo (for Liraglutide) 6 mg/ml once daily at a maximum dose of 1.8 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of liraglutide in the treatment of patients with idiopathic Parkinson's disease (PD).

DETAILED DESCRIPTION:
This single center, double-blind, placebo-controlled study will enroll 57 participants with a diagnosis of idiopathic PD. Subjects enrolled in the study will be randomized to receive once daily self-administered injections of liraglutide (1.2 or 1.8 mg, as tolerated) or placebo at the same dose range in a 2:1 study design.

Liraglutide has been approved by the Food and Drug Administration (FDA) to treat adults with Type 2 Diabetes (T2D) and to treat obesity, but it is considered investigational in this study, as it has not been approved for use in patients with PD. Liraglutide belongs to a class of medications able to stimulate receptors of glucagon-like peptide 1 (GLP-1), a naturally occurring peptide found throughout much of the brain and able to increase the incretin effect in patients with T2D, stimulating the release of insulin. Liraglutide can reduce systemic and brain insulin resistance, an abnormality that could help drive PD pathogenesis. Indeed, impaired insulin signaling in the brain can cause or exacerbate many brain pathologies and behavioral abnormalities seen in PD. Another GLP-1 agonist, named exenatide, has been evaluated in patients with PD, showing significant improvement of motor and cognitive symptoms. There is reason to believe that liraglutide may prove superior to exenatide in treating PD.

Eligible participants will be followed for up to 14 months and will be expected to complete 9 in-person visits and 2 telephone visits. The study will measure liraglutide effects on motor (assessed by changes in the MDS-UPDRS part III) and non-motor symptoms of PD (assessed by the NMSS and MDRS-2) after 52 weeks of treatment. The secondary outcomes include measures of the association between liraglutide's effects on peripheral insulin resistance, PD symptoms and safety. Collection of blood and urine samples will be obtained to monitor drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD according to the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria for at least 2 years
* Responsive to levodopa or dopaminergic treatment
* Male or female between 25 and 85 years of age at time of enrollment

  * Women of child-bearing potential (WOCBP) must agree to use a reliable method of contraception (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive, double barrier methods (such as condom plus diaphragm, condom plus spermicide foam, condom plus sponge), or intra-uterine devices) throughout the duration of the trial period and must have a negative serum pregnancy test at screening
  * Male patients with female partners who have child bearing potential must agree to use adequate contraception throughout the duration of the trial period
* Capacity to give informed consent
* Ability to self-administer, or to arrange a care partner to administer trial drug, to comply with trial protocol, and to attend necessary clinic visits off medication

Exclusion Criteria:

* Diagnosis or suspicion of other causes for Parkinsonism, including drug- or toxin-induced parkinsonism and other neurodegenerative conditions, including multiple system atrophy, progressive supranuclear palsy, Huntington's disease, Wilson's disease, or Alzheimer's disease
* Active treatment with anticholinergic medications (e.g., trihexyphenidyl, tricyclic antidepressants)
* Known abnormality on CT or MRI brain imaging considered to cause symptoms or signs of neurological dysfunction, or considered likely to compromise compliance with trial protocol
* Concurrent dementia defined by a score lower than 120 on the MADRS-2 and/or inability to complete scale per neuropsychologist discretion
* Concurrent severe depression defined by a score greater than 29 on the Beck Depression Inventory
* Prior intracerebral surgical intervention for PD, including deep brain stimulation, lesional surgery, growth factor administration, gene therapy, or cell transplant
* Already actively participating in a trial of a device, drug, or surgical treatment for PD, or trial participation within 30 days prior to the baseline visit
* Diagnosis of diabetes mellitus of any type, established historically or by:
* Fasting plasma glucose levels equal or above 126 mg/dl
* Hemoglobin A1c equal or above 6.5%
* Active treatment with oral antidiabetic medications
* History of severe cardiac disease (e.g., angina, myocardial infarction, or cardiac surgery) in the preceding year
* Significant systemic illness likely to result in deterioration of the patient's condition or, in the Investigator's opinion, affect the patient's safety during the study, including in particular:

  1. History of pancreatitis
  2. Personal or family history of medullary thyroid carcinoma
  3. History of multiple endocrine neoplasia syndrome type 2
  4. History of alcoholism
  5. Severe gastrointestinal disease, including gastroparesis
  6. Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within the last 90 days or chemotherapeutic agents for malignancy within the last 2 years
  7. Severe renal insufficiency (CrCl <30)
  8. Moderate or severe hepatic impairment
  9. Severe hypertriglyceridemia (triglycerides >500 mg/dl)
* Females who are pregnant or breast feeding
* Prior serious hypersensitivity reaction to Victoza or any of the product components 10) Body Mass Index <18.5

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tagliati, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Zhang L, Li Y, Li L, Melchiorsen JU, Rosenkilde M, Holscher C. The Novel Dual GLP-1/GIP Receptor Agonist DA-CH5 Is Superior to Single GLP-1 Receptor Agonists in the MPTP Model of Parkinson's Disease. J Parkinsons Dis. 2020;10(2):523-542. doi: 10.3233/JPD-191768. PMID 31958096

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 42 | 21
Completed | 33 | 18
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 42 | 21 | 63
Age, Customized [Number; unit: participants]
  40-49 years of age | 5 | 0 | 5
  50-59 years of age | 5 | 8 | 13
  60-69 years of age | 21 | 9 | 30
  70+ years of age | 11 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 29 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 40 | 21 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 42 | 19 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 21 | 63
Age of Onset [Mean (Standard Deviation); unit: years] — Age of Parkinson's disease symptom onset
  years | 58.7 (9.9) | 58.5 (7.4) | 58.6 (9.1)
Duration of Parkinson's Disease Symptoms [Mean (Standard Deviation); unit: years] | 5.3 (3.7) | 4.9 (3.2) | 5.1 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS Part III Motor Examination) During "OFF" Time From Baseline to the End of Double-Blind Maintenance Period
Description: The UPDRS Part III (motor symptoms sub-scale) Assessment consists of 17 items, measured on a 5-Point scale (0-Normal to 4-Severe), addressing speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability, and body bradykinesia. The participant's score is calculated as a sum of the scores of the 17 individual questions. This sum score ranges from 0 to 108. Higher scores denote greater disability.
  A participant has been considered "OFF" when he/she has been off L-dopa for greater than 12 hours. During "OFF" time, the participant will not report feeling the effects of their anti-Parkinson's medication. The participant recorded the exact time of L-dopa intake. Assessment was only conducted greater than 12 hours after dosing with the participant reportedly feeling "OFF."
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to 54 weeks)
Population: The Full Analysis Set (FAS) consisted of all subjects who were randomized, received at least 1 dose of study medication, had a valid Baseline primary efficacy measurement, and had at least 1 valid post-Baseline primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Full Analysis Set (Liraglutide-treated Subjects): Subjects receiving Liraglutide 6 mg/ml (Novo Nordisk A/S) self-administered subcutaneously once daily at a maximum dose of 1.8 mg after a 2-week titration schedule.
- Full Analysis Set (Placebo-treated Subjects): Subjects randomized to placebo self-administered matching placebo subcutaneously once daily according to the same schedule.
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | -2.3 (9.4) | -5.0 (7.1)

2. Primary Outcome: Change in the Non-Motor Symptoms Scale (NMSS) Total Score From Baseline to the End of the Double-Blind Maintenance Period
Description: The NMSS is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease. The NMSS measures severity and frequency of non-motor symptoms across nine dimensions (cardiovascular, sleep/fatigue, mood/apathy, perceptual problems/hallucinations, attention/memory, gastrointestinal, urinary, sexual function, and miscellaneous which includes pain, taste/smell, weight change, and excessive sweating). Higher scores indicate a higher burden of these symptoms on the patient.
  There are 30 items to be scored, and the item scores are calculated as the product of severity and frequency; the total score is obtained by summing the item scores. The NMSS total score ranges from 0 to 360 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: From Baseline (Week 0) to the End of Maintenance Period (up to Week 54)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | -5.5 (25.3) | 6.5 (21.3)

3. Primary Outcome: Change in the Mattis Dementia Rating Scale (DRS-2) From Baseline to the End of Double-Blind Maintenance Period
Description: The DRS-2 assesses individuals in five areas resulting in five sub-scale scores. These scores are used to determine the overall score and level of cognitive functioning ability. The five areas include:
  Attention - measured using eight items Construction - measured using six items Conceptualization - measured using six items Initiation/Preservation - measured using eleven items Memory - measured using five items Higher raw scores indicate better cognitive status, with scores ranging from 0 to 144. Normative data in healthy subjects range from 137 to 144.
Time Frame: From Baseline (Week 0) to the end of Maintenance Period (up to 54 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Full Analysis Set (Liraglutide-treated Subjects): Subjects receiving Liraglutide 6 mg/ml (Novo Nordisk A/S) self-administered subcutaneously once daily at a maximum dose of 1.8 mg after a 2 week titration schedule.
- Full Analysis Set (Placebo-treated Subjects): Subjects randomized to receiving Placebo self-administered matching placebo subcutaneously once daily according to the same schedule.
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | 1.4 (9.3) | -0.3 (9.1)

4. Secondary Outcome: Change in the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Index From Baseline to the End of Maintenance Period
Description: Peripheral insulin resistance was assessed using the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Index. The HOMA-IR tool is a validated, non-invasive tool to assess the relationship between glucose and insulin. A score less than 1 means indicates insulin-sensitivity (Optimal). Greater than 1.9 indicates early insulin resistance, and a score greater than 2.9 indicates significant insulin resistance.
  An increase in one's HOMA-IR score may indicate increased insulin resistance.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to 54 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | 0.1 (1.1) | 0.3 (0.8)

5. Secondary Outcome: Change in the Unified Parkinson's Disease Rating Scale Total Score From Baseline to the End of Double-Blind Maintenance Period
Description: Total UPDRS Score (Parts I, II, III, and IV; administered in the ON condition) Change from Baseline to End of Maintenance Period.
  UPDRS I evaluation of mentation, behavior, and mood UPDRS II self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food UPDRS III clinician-scored monitored motor evaluation UPDRS IV evaluation of complications in therapy and motor fluctuations, including OFF time and dyskinesia
  The UPDRS I, II, III, and IV scores and subscores are calculated as the sum of all individual items.
  Subscales have 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe
  The final cumulative score will range from 0 (no disability) to 260 (total disability). A decrease in the mean indicates global improvement in the UPDRS score.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to 54 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | -4.9 (12.7) | 2.3 (10.4)

6. Secondary Outcome: Change in The Parkinson's Disease Questionnaire (PDQ-39) From Baseline to the End of Double-Blind Maintenance Period
Description: The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item patient-reported rating scale that measures Parkinson's disease-specific health related quality of life.
  It covers 8 areas: mobility, activities of daily living (ADL), emotional well-being, stigma, social support, cognition, communication and bodily discomfort.
  Lower scores indicate better health related quality of life. PDQ-39 total scores range from 0 to 800. The total score can be summarised into the PDQ-39 summary index score (range of scores 0 to 100). A mean change in the PDQ-39 summary index score of about 1.6 points relates to feeling 'a little worse' and is likely to represent a clinically important difference.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to 54 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Full Analysis Set (Placebo-treated Subjects): Subjects receiving Placebo self-administered matching placebo subcutaneously once daily according to the same schedule.
Arm/Group | Full Analysis Set (Liraglutide-treated Subjects) | Full Analysis Set (Placebo-treated Subjects)
Number analyzed (Participants) | 33 | 18
units on a scale | -2.5 (9.9) | 11.2 (14.0)

ADVERSE EVENTS:
Time Frame: Adverse Event collection commenced upon signing of consent at Screening and occurred at Baseline Week 1, Week 2, Week 6, Week 14, Week 28, Week 38, Week 54, and at follow-up Week 58.
Groups:
- Liraglutide: Liraglutide 6 mg/ml (Novo Nordisk A/S) self-administered subcutaneously once daily at a maximum dose of 1.8 mg after a 2 week titration schedule.
  Liraglutide: Liraglutide 6 mg/ml once daily at a maximum dose of 1.8 mg
- Placebo: Matching Placebo self-administered subcutaneously once daily according to the same schedule.
  Placebo: Placebo (for Liraglutide) 6 mg/ml once daily at a maximum dose of 1.8 mg
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/21
Serious Adverse Events (participants affected / at risk) | 9/42 | 2/21
Other Adverse Events (participants affected / at risk) | 42/42 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liraglutide (N=42) | Placebo (N=21)
Fall/Admission for Fall (Injury, poisoning and procedural complications) | 2 | 0
Urinary Tract Infection (UTI)/Admission for UTI (Renal and urinary disorders) | 1 | 0
Dizziness/Admission for Dizziness (Nervous system disorders) | 1 | 0
Hospital Admission for Averted Stroke (Vascular disorders) | 0 | 1 — Subject reported right-sided facial numbness, dizziness, clumsiness. He subsequently went to the hospital. Imaging was negative and the subject received tPA. Follow-up imaging revealed no infarct or bleed.
Worsening Urinary Retention (Renal and urinary disorders) | 1 | 0
Hospital Admission for Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Prostate Cancer (Renal and urinary disorders) | 1 | 1
Squamous Cell Carcinoma of Cervix (Reproductive system and breast disorders) | 1 | 0
Invasive Lobular Carcinoma (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=42) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 24 (31) | 3 (4)
Loss of Appetite (Metabolism and nutrition disorders) | 26 (26) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 12 (16) | 3 (3)
Injection Site Reaction (General disorders) | 10 (10) | 3 (4) — General Disorders and Administrative Site Conditions
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (8) | 2 (2)
Other Pain (Nervous system disorders) | 7 (7) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 2 (2)
Sleep Disorder (Nervous system disorders) | 4 (4) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0)
Worsening Off Time (Nervous system disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
A single-center trial may prevent broad generalization of the results, and reduced the variability in data collection. There was a lack of diversity; a vast majority of study subjects were Caucasian. We did not collect cerebrospinal fluid (CSF) data, which may limit data interpretation. The lack of a video-recorded MDS-UPDRS prevented an independent review of motor scores that could have ruled out observer bias as the explanation for the recorded placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02953665/Prot_SAP_000.pdf